CLINICAL TRIAL: NCT01655823
Title: A Randomized, Double-Blind, Dose-Finding, Placebo Controlled, Phase II Multicenter Study of Tetrodotoxin in the Treatment of Chemotherapy Induced Neuropathic Pain
Brief Title: The Purpose of This Study is to Determine if Tetrodotoxin (TTX) is Effective in the Treatment of Pain Resulting From Chemotherapy Treatment
Acronym: TTX-CINP-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis completed and decided to terminate and proceed to Phase 3 trial.
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTX-CINP-201
Record Dates: First submitted 2012-07-19; First posted 2012-08-02 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pain; Peripheral Neuropathy; Neuropathic Pain
Keywords: Pain; Puffer fish; Tetrodotoxin; TTX; Neuropathy; Chemotherapy; WEX Pharmaceuticals
MeSH Terms: conditions — Pain; Peripheral Nervous System Diseases; Neuralgia | interventions — Injections; Tetrodotoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (twice daily) (Placebo Comparator): Placebo for injection (1 ml volume), twice a day for four consecutive days.
  Interventions: Drug: Placebo
- Low dose Tetrodotoxin (twice daily) (Experimental): Low dose Tetrodotoxin injectable (1 ml volume), twice a day for four consecutive days.
  Interventions: Drug: Tetrodotoxin
- Mid-range dose of Tetrodotoxin (twice daily) (Experimental): Mid-range dose Tetrodotoxin injectable (1 ml volume), twice a day for four consecutive days.
  Interventions: Drug: Tetrodotoxin
- Max dose Tetrodotoxin (once daily) (Experimental): Max dose Tetrodotoxin injectable (1 ml volume), once a day in the morning for four consecutive days and Placebo for injection (1 ml volume), once a day in the afternoon for four consecutive days. Total of 4 treatment days.
  Interventions: Drug: Placebo; Drug: Tetrodotoxin
- Max dose Tetrodotoxin (twice daily) (Experimental): Max dose Tetrodotoxin injectable (1 ml volume), twice a day for four consecutive days.
  Interventions: Drug: Tetrodotoxin

INTERVENTIONS:
Drug: Placebo — Sham treatment acting as control arm
  Other Names: placebo for injection
  Arms: Max dose Tetrodotoxin (once daily); Placebo (twice daily)
Drug: Tetrodotoxin — Comparison of different dosages of Tetrodotoxin
  Other Names: TTX for injection
  Arms: Low dose Tetrodotoxin (twice daily); Max dose Tetrodotoxin (once daily); Max dose Tetrodotoxin (twice daily); Mid-range dose of Tetrodotoxin (twice daily)

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a major dose-limiting side effect of many chemotherapeutic agents including vincristine, paclitaxel, cisplatin, oxaliplatin, bortezomib and ixabepilone. Chemotherapy-induced peripheral neuropathy commonly occurs in greater than 40% of patients. To improve the peripheral neuropathy, the chemotherapy dosing is often either decreased or discontinued potentially affecting tumor responsiveness, prognosis, and survival.

There is an unmet medical need for treatment of cancer patients with chemotherapy induced neuropathic pain (CINP) and the proposed study will investigate the efficacy and safety of multiple dose levels of tetrodotoxin (TTX) versus placebo in moderate to severe neuropathic pain caused by chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* If female, not of childbearing potential.
* Patients with documented neuropathic pain
* Cancer Patients who have completed a chemotherapy regimen which included taxanes or platinums (or both) and have no evidence actively progressive disease. Concurrent hormonal therapies are allowed
* Patients with stable moderate to severe neuropathic pain
* Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Patients who are able to complete the study-related questionnaires independently in either English or Spanish.

Exclusion Criteria:

* History of peripheral neuropathy attributed to any cause other than chemotherapy.
* Patients receiving any concurrent agents known to cause peripheral neuropathy within 30 days of Randomization.
* Current use of other therapy (ies), including "alternative" therapies, for treatment of peripheral neuropathy within 30 days of Randomization (with the exception of protocol allowed concurrent medications).
* Patients who used controlled release opioids within seven days of baseline period or who expect to use controlled release opioids at any time from baseline to end of study.
* Patients with abnormal kidney function.
* Patients with bone metastases.
* Patients scheduled for treatment for their cancer with chemotherapy or radiotherapy between screening and the end of study visit.
* Current use of lidocaine and other types of antiarrhythmic drugs within 30 days of Randomization.
* Current use of scopolamine and acetylcholinesterase-inhibiting drugs such as physostigmine within 30 days of Randomization.
* Current cause of Chemotherapy Induced Neuropathic Pain attributed to Velcade (Bortezomib) or vinca alkaloids or analogues such as vincristine, vinblasine, vinorelbine and vindesine.
* Current use of tricyclic antidepressant medication, anticonvulsants and monoamine oxidase inhibitors.
* Patients with current uncontrolled asthma or lung disease.
* Patients with significant heart disease.
* Use of an investigational agent within 30 days prior to screening or is scheduled to receive an investigational drug other than TTX during the course of the study.
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Goldlust, MD, Principal Investigator — Hackensack University
Locations (23):
- United States (23):
  - Lalita Pandit, Fountain Valley, California
  - Robert Moss, Fountain Valley, California
  - Alliance Research Centers, Laguna Hills, California
  - Global Research Management, Los Angeles, California
  - Innovative Clinical Research, Los Angeles, California
  - El Camino Cancer Center, Mountain View, California
  - Pacific Cancer Care, Salinas, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Axcess Medical Research, Wellington, Florida
  - Cancer Center of Middle Georgia, Dublin, Georgia
  - Cancer Center of Kansas, Wichita, Kansas
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - St. Louis Cancer Care, Bridgeton, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Institute of Pain Research, Oklahoma City, Oklahoma
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo (Twice Daily) | Low Dose Tetrodotoxin (Twice Daily) | Mid-range Dose of Tetrodotoxin (Twice Daily) | Max Dose Tetrodotoxin (Once Daily) | Max Dose Tetrodotoxin (Twice Daily)
Started | 25 | 25 | 24 | 25 | 26
Completed | 25 | 23 | 24 | 24 | 25
Not Completed | 0 | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Twice Daily) | Low Dose Tetrodotoxin (Twice Daily) | Mid-range Dose of Tetrodotoxin (Twice Daily) | Max Dose Tetrodotoxin (Once Daily) | Max Dose Tetrodotoxin (Twice Daily) | Total
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 26 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.3) | 59.1 (10.29) | 61.4 (10.01) | 60.4 (10.28) | 60.6 (11.05) | 60.1 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 15 | 16 | 77
  Male | 10 | 9 | 9 | 10 | 10 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 24 | 25 | 26 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient Reported Outcome for Pain at Day 22 to Day 28.
Description: The primary efficacy endpoint for Part I was the change from baseline in weekly average NPRS scores at 22 to 28 days after treatment. Baseline was defined as the average of NPRS scores for the last 7 days prior to dosing. Pain was assessed using a Numerical Pain Rating Scale (NPRS) with a range of 0 (no pain) to 10 (extreme pain).
Time Frame: Day 22 to Day 28
Population: ITT
Measure: Mean (Standard Deviation); unit: 11 point units on a scale
Arm/Group | Placebo (Twice Daily) | Low Dose Tetrodotoxin (Twice Daily) | Mid-range Dose of Tetrodotoxin (Twice Daily) | Max Dose Tetrodotoxin (Once Daily) | Max Dose Tetrodotoxin (Twice Daily)
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 26
11 point units on a scale
  Baseline | 6.662 (1.4832) | 6.285 (1.3312) | 7.012 (1.3706) | 6.240 (1.1743) | 6.255 (1.3561)
  Mean Scores for Days 22-28 | 5.323 (2.2765) | 5.005 (2.0451) | 5.987 (2.2531) | 4.566 (2.4931) | 4.749 (1.7701)
  Change from Baseline in Mean Scores for Days 22-28 | -1.339 (2.0681) | -1.269 (1.3959) | -1.052 (1.5742) | -1.682 (2.3231) | -1.529 (1.8203)

ADVERSE EVENTS:
Arm/Group | Placebo (Twice Daily) | Low Dose Tetrodotoxin (Twice Daily) | Mid-range Dose of Tetrodotoxin (Twice Daily) | Max Dose Tetrodotoxin (Once Daily) | Max Dose Tetrodotoxin (Twice Daily)
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25 | 1/24 | 0/25 | 1/26
Other Adverse Events (participants affected / at risk) | 18/25 | 21/25 | 22/24 | 20/25 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Twice Daily) (N=25) | Low Dose Tetrodotoxin (Twice Daily) (N=25) | Mid-range Dose of Tetrodotoxin (Twice Daily) (N=24) | Max Dose Tetrodotoxin (Once Daily) (N=25) | Max Dose Tetrodotoxin (Twice Daily) (N=26)
Metastatic carcinoma of bladder and Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Twice Daily) (N=25) | Low Dose Tetrodotoxin (Twice Daily) (N=25) | Mid-range Dose of Tetrodotoxin (Twice Daily) (N=24) | Max Dose Tetrodotoxin (Once Daily) (N=25) | Max Dose Tetrodotoxin (Twice Daily) (N=26)
Paraesthesia (Nervous system disorders) | 6 | 5 | 7 | 5 | 10
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 1 | 2 | 1
headache (Nervous system disorders) | 5 | 6 | 3 | 1 | 9
dizziness (Nervous system disorders) | 5 | 3 | 4 | 3 | 8
Paraesthesia Oral (Nervous system disorders) | 3 | 4 | 9 | 10 | 11
Hypoaesthesia Oral (Nervous system disorders) | 3 | 5 | 7 | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less